CLINICAL TRIAL: NCT05268432
Title: Development, Intraoperative Demonstration and Visualization of Surgical Assistance Functions
Acronym: IDEMONSTRATE
Status: Recruiting | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Other Study IDs: VTG-09
Record Dates: First submitted 2022-02-07; First posted 2022-03-07 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Abdominal Surgery
Keywords: Surgical data science; computer vision
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Surgery with intraoperative imaging — laparoscopic, robot-assisted or other intraoperative imaging (ultrasound, CT, MRI)

SUMMARY:
The aim of the planned study is the development of surgical assistance functions on the basis of clinical routine data and the evaluation of the technical feasibility of an intraoperative demonstration and visualization of such assistance functions in visceral surgery. Furthermore, this trial aims to provide preliminary data on the clinical outcome of such assistance systems.

DETAILED DESCRIPTION:
The aim of the clinical trial is to create the conditions for the comprehensive scientific use of new technologies such as augmented and virtual reality, computer-aided navigation and robotics in surgery in order to use these technologies in the future for improved surgical therapy for the benefit of the patient and to support the treating surgical team. The IDEMONSTRATE study is divided into two study parts: the development of a surgical assistance function based on routinely collected clinical (image) data that displays the position of anatomical structures (e.g. blood vessels, organs, tumors) in real time and the technical evaluation of this assistance system in the clinical environment.

For the development of the surgical assistance function, data routinely collected as part of surgical inpatient treatment will be used. For research purposes (and explicitly not to prepare for approval as a medical device), a surgical assistance function is to be developed from this that displays the position of anatomical structures in real time during visceral surgical interventions. This system will then be evaluated in the second part of the study with regard to its technical feasibility and medical relevance.

For the evaluation of the developed assistance function in the context of clinical treatment, the patients and the staff involved will be informed separately. All patients who are eligible for inclusion in the evaluating part of the study are fully capable of giving their consent. All doctors who will take part in the evaluation of the developed algorithm in a clinical context are specialists in general or visceral surgery; these doctors are informed in detail about the risks and sources of error in the context of the application before the developed algorithm and the associated assistance function is used. The evaluation of the developed assistance function takes place exclusively in the context of planned interventions, not in emergency situations.

ELIGIBILITY:
Inclusion Criteria:

* Indication for surgery using a laparoscopic or open surgical camera, a surgical robot (e.g., DaVinci system), or an intraoperative imaging modality (e.g. sonography, intraoperative CT)
* Patient understands German

Exclusion Criteria:

* Lack of ability to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll patients undergoing surgery using a laparoscopic or open surgical camera, a surgical robot (e.g. DaVinci®), or intraoperative imaging technology (e.g. ultrasound, CT).
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-05-19 (Actual); Primary Completion 2050-12-31 (Estimated); Study Completion 2050-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of intraoperative technical errors of the applied assistance system | during surgery
  Major technical errors: system crash, calculation latency > 1 second, Image distortions

SECONDARY OUTCOMES:
Evaluation of surgical skills | during surgery
  The IDEMONSTRATE skill assessment scale v1.0 will be used to rate surgical skill on a scale from 1 to 5, with higher scores indicating higher skill levels.
Display accuracy of guidance functions | during surgery
  The IDEMONSTRATE display accuracy scale v1.0 will be used to rate display accuracy on a scale from 1 to 5, with higher scores indicating better display accuracy.
Operating time [min] | during surgery
  Time from skin incision until placement of last skin staple/suture
Duration of postoperative hospital stay [days] | At day of discharge, assessed up to 90 days
  Postoperative day 1 until day of discharge
Duration of postoperative intermediate/intensive care unit stay [days] | At day of discharge, assessed up to 90 days
  Postoperative day 1 until day of discharge
Frequency of peri-operative morbidity after resection | At day of discharge, assessed up to 90 days
  Frequency of peri-operative complications after surgery
Kind of peri-operative morbidity after resection | At day of discharge, assessed up to 90 days
  Kind of peri-operative complications after surgery
Assessment of usability of guidance system | 48 hours after surgery
  Surgeon questionnaire, the questionnaire qualitatively assesses nine items, each item scoring from "not at all" to "very much", evaluated individually

CONTACTS AND LOCATIONS:
Overall Officials: Marius Distler, Prof. Dr., Principal Investigator — Technical University Dresden
Locations (1):
- Department of Gastrointestinal-, Thoracic and Vascular Surgery University Hospital Carl Gustav Carus Technische Universität Dresden, Dresden, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No
Following publication of study results, de-identified patient data may be made available upon reasonable request